CLINICAL TRIAL: NCT01615562
Title: Endothelial Dysfunction in Adolescents and Women With Polycystic Ovary Syndrome (PCOS)
Brief Title: Blood Vessel Function in Adolescents and Women With Polycystic Ovary Syndrome
Status: Terminated | Type: Observational
Why Stopped: Difficulty in enrolling suitable subjects
Sponsor: Virginia Commonwealth University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: U54HD034449- Wickham Pilot; U54HD034449 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Last update posted 2015-12-14 (Estimated); Status verified 2015-12

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: Polycystic Ovary Syndrome; PCOS; Infertility
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum and plasma for analysis of hormones
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- PCOS adolescents: Post-menarchal females ages 14-17 with and without PCOS (15 each group for a total of 30 subjects).
- PCOS women: Women ages 18-40 with and without PCOS (15 each group for a total of 30 subjects).

SUMMARY:
The purpose of this study is to determine if changes in blood vessel health lead to the menstrual irregularities that women with PCOS experience. This research study will help determine if women with PCOS have early changes in their blood vessels called "endothelial dysfunction," and if the number of progenitor cells (cells that in a healthy person repair blood vessel damage) are related to these blood vessel changes. To do so, we will compare ultrasound (soundwave) pictures of a large blood vessel in the arm and the results of blood tests between women with PCOS and other healthy women with normal menstrual periods.

DETAILED DESCRIPTION:
Overview:

Although adult women with PCOS demonstrate evidence of endothelial dysfunction, little is known regarding alterations in the number of pro-inflammatory monocytes, CEC, CPC, and ECFC (endothelial injury/repair profile) among affected women. For many women, the clinical manifestations of PCOS emerge during adolescence. Based on studies documenting the increased prevalence of MetS and inflammatory markers in adolescent girls with PCOS, and non-invasive studies documenting the presence of endothelial dysfunction in children with traditional cardiovascular risk factors, it is likely adolescent girls with PCOS already manifest evidence of early vascular dysfunction, which may in turn impair follicular development and contribute to the development of infertility.

Consequently, we hypothesize that perturbations in the balance between circulating inflammatory and progenitor cells contribute to the endothelial dysfunction observed in adult women with PCOS. Specifically, we anticipate that PCOS women will manifest greater evidence of vascular injury (increased numbers of inflammatory monocytes, CEC, and ECFC) and impaired endothelial repair (decreased levels of CPC) compared with control women. Moreover, we propose that, in adolescent girls with PCOS, endothelial dysfunction and corresponding alterations in the endothelial injury/repair profile are already present.

Specific Aim 1: Determine if the endothelial injury/repair profile (inflammatory monocytes, CEC, CPC, and ECFC) assessed by flow cytometry (PFC) and endothelial function (assessed by flow-mediated vasodilation (FMD) of the brachial artery) are altered in treatment-naïve adult (18-40 years of age) women with PCOS (n=15) compared with age and body mass index (BMI)-matched control women (n=15).

Specific Aim 2: Determine if the endothelial injury/repair profile assessed by PFC, AGE levels, and endothelial function (assessed by FMD of the brachial artery) are altered in treatment-naïve adolescents (14-17 years of age) with PCOS (n=15) compared with age and BMI-Z-score-matched control girls (n=15).

Specific Aim 3: Determine if observed alterations in the endothelial injury/repair profile (pro-inflammatory monocytes, CEC, CPC and ECFC) or levels of AGE correlate with endothelial function (assessed by FMD of the brachial artery) in adolescent and adult women with (n=30) and without PCOS (n=30), and whether androgens, insulin resistance, or other cardiovascular risk factors influence these relationships.

This is a cross-sectional study design involving 30 post-menarchal adolescents and 30 adult female subjects. Specifically, the adolescent population will include 15 treatment-naïve adolescent females (ages 14-17 years) with PCOS and 15 age- and BMI-percentile-matched control adolescent subjects. Similarly, the adult study population will include 15 treatment-naïve adult females (ages 18-40 years) with PCOS and 15 age- and BMI-matched control women. All study procedures will be conducted at the Clinical Research Services Unit (CRSU) at Virginia Commonwealth University (VCU) during a single visit (~3.5 hrs).

CRSU Visit:

Subjects will be admitted to the CRSU after a 12-hour overnight fast. Subjects will also be instructed to refrain from vigorous physical activity for 24 hours prior to the visit. All participants will undergo a detailed medical history (including a menstrual history) and a complete physical examination (including assessments of Tanner Staging for breast and pubic hair development). Hirsutism will be assessed using the modified Ferriman-Gallwey scoring system.

At the study visit, the following anthropometric measurements with be performed on all subjects:

* Blood pressure obtained in left arm - 3 readings at 5 minute intervals
* Pulse
* Temperature
* Height (2 measurements)
* Weight (2 measurements)
* Waist/umbilicus/hip circumference measurements (2 measurements)
* Bioimpedence

At the study visit a resting electrocardiogram (ECG) will be obtained for all subjects.

At the study visit, the following labs will be obtained on all subjects:

* Comprehensive metabolic panel
* Lipid panel
* Urine pregnancy
* TSH*
* Prolactin*
* 17-hydroxyprogesterone*
* Testosterone* *These analyses are to be performed only when additional eligibility screening is needed and only at PI request.

All subjects will undergo measurement of brachial artery flow-mediated vasodilation (FMD). FMD testing will be performed by the PI or Co-Investigator in the CRSU Peripheral Vascular Lab with the assistance of a trained technician using an ultrasound peripheral vascular imaging system. Adult subjects only will also undergo brachial artery reactivity testing for the assessment of non-endothelial dependent (NED) vessel dilation following the administration of nitroglycerin. NED testing will be performed following a rest period of at least 15 minutes from completion of the FMD testing. 400 μg of nitroglycerin will be administered sublingually, and images will be recorded for at least 3 minutes following the administration of nitroglycerin.

Following the FMD testing (allow 30 minute interval), all subjects are to undergo a 2-hour 75 g oral glucose tolerance test.

• Samples collected at baseline (-15 and 0) and 30 minute intervals for glucose, insulin

ELIGIBILITY:
Inclusion Criteria:

* PCOS as defined by NIH/NICHD criteria: 1) oligo- or amenorrhea (≤8 menstrual periods annually, persisting 2 years post menarche); 2) biochemical hyperandrogenism(HA), i.e.,elevated total or free testosterone concentration and/or clinical evidence of HA (defined as the presence of hirsutism); and 3) exclusion of secondary causes of ovulatory dysfunction and HA (including hyperprolactinemia, thyroid dysfunction, non-classical congenital adrenal hyperplasia (NCAH) due to 21-hydroxylase deficiency, Cushing syndrome, androgen secreting neoplasms, and androgenic/anabolic drug use).
* Inclusion criteria for adolescent and adult control subjects will include 1) normal menstrual periods (defined as regular cycles between 22-36 days in length); 2) normal serum androgens (total/free testosterone and dehydroepiandrosterone-sulfate [DHEA-S]); and 3) absence of clinical evidence of hyperandrogenism. Additionally, adolescent controls must be 2 years post menarche.

Exclusion Criteria:

* Diabetes mellitus
* Underlying endocrine, neurologic, and/or genetic syndromes leading to obesity
* Congenital heart disease or abnormal resting ECG
* Renal or hepatic disease
* History of rheumatologic disorders or malignancy
* Use of medications or dietary supplements known to affect insulin sensitivity (i.e. metformin, corticosteroids, and oral contraceptive pills), blood pressure, or cholesterol within 3 months of study participation
* Investigation drug use within 3 months of study participation
* Pregnancy
* Current tobacco use

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Specifically the study will enroll: 15 treatment-naïve adolescents with PCOS; 15 age- and BMI Z-score matched adolescent controls without PCOS; 15 adult treatment-naïve women with PCOS; and 15 age- and BMI-matched adult women without PCOS. Subject race/ethnicity is not a specific inclusion/exclusion criterion for this study.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2011-12; Primary Completion 2014-04 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Peripheral vascular imaging via ultrasonography during brachial artery flow-mediated vasodilation (FMD) | ~ 30 minutes
  A blood pressure cuff is placed on right forearm. A 7-12MHz linear array ultrasound transducer is placed on upper arm. 2-D and Doppler images are acquired. Forearm cuff is inflated to ~ 50 mmHg above resting systolic blood pressure (max 300 mmHg) for 4.5 minutes, then deflated. Blood flow velocity via Doppler is recorded for 15 seconds; 2D-images of the brachial artery are collected for 3 minutes. Brachial artery diameter is measured at end diastole (R-wave on ECG).FMD is determined: %FMD=(LDp-LDb)/LDbx100, where LDp=luminal diameter after inflation and LDb=luminal diameter at baseline

SECONDARY OUTCOMES:
FMD with non-endothelial dependent (NED) vessel dilation | ~30 minutes
  NED testing will be performed following a rest period of at least 15 minutes from completion of the FMD testing. For NED testing, a second baseline and 2D image and Doppler signal will be performed as previously outlined. Following repeat baseline imaging, 400 μg of nitroglycerin will be administered sublingually, and images will be recorded for at least 3 minutes following the administration of nitroglycerin. Only adult subjects will undergo NED.

CONTACTS AND LOCATIONS:
Overall Officials: Edmond Wickham, MD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Virginia Commonwealth University, Richmond, Virginia, United States

REFERENCES:
- See also: VCU PCOS Research Site — http://www.vcu.edu/pcos/research.html